CLINICAL TRIAL: NCT04282928
Title: A Singlecenter, Randomized, Open Lable, Intervention Controlled Clinical Study on the Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells for the Treatment of Severe Viral Pneumonia
Brief Title: Efficacy and Safety of Umbilical Cord Mesenchymal Stem Cells for the Treatment of Severe Viral Pneumonian
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC.D（BG）.013.02.0
Record Dates: First submitted 2020-02-13; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Severe Pneumonia
Keywords: Umbilical Cord Mesenchymal Stem Cells; Severe viral Pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine treatment group (Active Comparator): Participants will receive the treatment according to the treatment principle of severe and critical cases in "Influenza diagnosis and treatment plan (2019 version)"
  Interventions: Procedure: Routine treatment
- HUC-MSCs adjuvant Group (Experimental): Participants will receive intravenous infusion of definitive HUC-MSCs (1×10^6 cells/Kg × body weight(kg), which was selected by immunomodulatory assay through coculture with BV2 cell) on the basis of the routine treatment.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells; Procedure: Routine treatment

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — Definitive Human umbilical cord mesenchymal stem cells selected by immunomodulatory assay through coculture with BV2 cell
  Arms: HUC-MSCs adjuvant Group
Procedure: Routine treatment — According to"Influenza diagnosis and treatment plan (2019 version)"

SUMMARY:
The purpose of this clinical study is to answer the questions:

1. Is the proposed intervention safe?
2. Is the proposed intervention effective in improving the health of subjects with severe viral pneumonia？

DETAILED DESCRIPTION:
Viral pneumonia is an acute respiratory infectious disease caused by respiratory viruses. It is mainly caused by the invasion of respiratory viruses such as influenza virus and adenovirus into the lower respiratory tract. Every winter and spring is the epidemic season. Influenza virus and adenovirus have high infectivity and pathogenicity. The rapid progress of some patients may be caused by acute respiratory distress syndrome (ARDS) or multiple organ dysfunction And died of complications. The fatality rate of severe patients is 9.8% - 60%. Most of the dead cases were the elderly and the patients with basic diseases. In addition to the complications, the main cause of death is ARDS caused by virus infection, on the other hand, the basic immune function of the elderly is poor, so it is difficult to form an effective antiviral response in response to virus infection. The direct destruction of the alveolar epithelial barrier and the systemic inflammatory response induced by the infection, namely, the destruction of the alveolar capillary barrier by the inflammatory waterfall, are the important pathogenesis of ARDS. How to effectively regulate the inflammatory response, prevent the inflammatory exudation and edema of the lungs, improve oxygenation, and reduce organ damage; at the same time, how to effectively improve the basic immune function and enhance the anti-virus immune response of such patients, has become the key to the success of the treatment of patients with severe viral pneumonia.

Umbilical cord mesenchymal stem cells (UC-MSCs) can differentiate into the different germ layers and play an important role in immune regulation and damage repair regulation. Clinical trials have shown that MSC is safe and effective in the treatment of acute lung injury and pulmonary fibrosis, and it can improve the immune function of patients with viral infectious diseases. Hence, intravenous infusion of HUC-MSCs is attractive therapy against severe viral pneumonia.

This is a randomized, singlecenter, open lable, intervention controlled clinical trial. The participants (n = 40) will be randomly distributed into two groups. The routine treatment group (n = 20) will receive the treatment according to "Influenza diagnosis and treatment plan (2019 version)", the HUC-MSCs adjuvant Group (n = 20) will receive intravenous infusion of definitive HUC-MSCs (1×10^6 cells/Kg × body weight(kg), which was selected by immunomodulatory assay through coculture with BV2 cell) on the basis of the routine treatment once at day 1 after joining. Follow-up duration is 90 days. The difference of 90 day mortality and average length of stay between the two groups will be observed and recorded. The changes of inflammatory index, viral load, oxygenation index and pulmonary imaging will be monitored at different time points after treatment in the two groups. The serious adverse events (SAEs) and adverse events (AEs) will be observed during the period.

The intent of this study is to explore the efficacy of HUC-MSCs in the treatment of severe viral pneumonia through improving the antiviral immune response of patients, reduce the lung inflammatory damage caused by the virus and the pulmonary interstitial fibrosis after the injury, and finally achieve the goal of reducing the mortality and improving the prognosis of severe patients, and to evaluate the safety.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18-75 years old (inclusive), and the gender is not limited;
2. According to the diagnosis standard of viral pneumonia in the influenza diagnosis and treatment plan (2019 version), patients with severe viral pneumonia were diagnosed.
3. Diagnostic criteria of viral pneumonia: with clinical manifestations of influenza, with one or more of the following pathogenic test results positive: 1) influenza virus nucleic acid test positive. 2) influenza antigen was positive. 3) the culture of influenza virus was positive. 4) the level of influenza virus specific IgG antibody in the acute and recovery serum was 4 times or more higher. Diagnosis criteria of severe viral pneumonia: the confirmed patients meet any of the following criteria: 1) continuous high fever for more than 3 days, accompanied by severe cough, expectoration, blood sputum, or chest pain; 2) rapid respiratory rate, dyspnea, cyanosis of mouth and lips; 3) mental changes: slow response, drowsiness, agitation, convulsion, etc.; 4) severe vomiting, diarrhea, dehydration; 5) pneumonia; 6 ）7. Other clinical conditions requiring hospitalization
4. 20kg / m2 ≤ BMI ≤ 30 kg / m2;
5. Volunteer to participate in the clinical study and sign the written informed consent.

Exclusion Criteria:

1. Long term use of immunosuppressive drugs or organ transplantation;
2. T lymphocyte abnormality (the use of allogeneic may be considered, according to the clinical opinion), HIV positive;
3. High allergic constitution or severe allergic history, especially IL-2 allergic history;
4. Pregnant and lactating women;
5. Patients with a history of serious autoimmune diseases; those who are allergic to all biological agents in the treatment, such as IL-2;
6. Patients with serious complications: Patients with chronic cardiac insufficiency (NYHA cardiac function grade IV), chronic renal insufficiency (CKD stage 4 or above), chronic liver insufficiency (child Pugh score > 12), and patients with malignant tumors.
7. There are other situations that the researcher thinks are not suitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
mortality | 90 day
  The difference of 90 day mortality between the two groups will be observed and recorded
average length of stay | 90 day
  The difference of average length of stay between the two groups will be observed and recorded

SECONDARY OUTCOMES:
Changes of inflammatory index - the number of leukocyte or lymphocyte | Day 0, Day 1，Day 3，Day 7，Day 14，Day 30，Day 60，Day 90
  Before the infusion of UC MSCs and on the 1st, 3rd, 7th, 14th, 30th, 60th and 90th day after the infusion, the peripheral blood of the patients will be collected to detect the number of leukocyte (10^9/L) or lymphocyte (10^9/L).
Changes of inflammatory index - the percentage of lymphocytes | Day 0, Day 1，Day 3，Day 7，Day 14，Day 30，Day 60，Day 90
  Before the infusion of UC MSCs and on the 1st, 3rd, 7th, 14th, 30th, 60th and 90th day after the infusion, the peripheral blood of the patients will be collected to detect the percentage of lymphocytes(%).
Changes of inflammatory index - cytokines | Day 0, Day 1，Day 3，Day 7，Day 14，Day 30，Day 60，Day 90
  Before the infusion of UC MSCs and on the 1st, 3rd, 7th, 14th, 30th, 60th and 90th day after the infusion, the peripheral blood serum of the patients will be collected to detect the level of CRP, SAA, ESR, PCT and IL-6 (μg/L).
Changes of oxygenation index | Day 0, Day 1，Day 3，Day 7，Day 14，Day 30，Day 60，Day 90
  Before the infusion of UC MSCs and on the 1st, 3rd, 7th, 14th, 30th, 60th and 90th day after the infusion, the arterial blood of the patients will be analyzed and the oxygenation index (mmHg) will be calculated according to the oxygen concentration of the patients. The change trend of the oxygenation index will be observed.
Throat swab/blood viral load | Day 0, Day 1，Day 3，Day 7，Day 14，Day 30，Day 60，Day 90
  Before the infusion of UC MSCs and on the 1st, 3rd, 7th, 14th, 30th, 60th and 90th days after the infusion, the throat swabs and peripheral blood were collected respectively. The RNA copies of the virus will be detected by RT-PCR. The change trend of the viral load in the throat swabs/peripheral blood of the patients in each group will be observed after the treatment with different regimens, and the difference of the viral load between different groups will be compared
Chest imaging outcome | Day 0, Day 7, Day 30, Day 90
  Two senior (associate chief physician and above) respiratory radiologists read the films independently. The chest CT images of the two groups will be evaluated before UC-MSCs infusion and on the 7th, 30th and 90th day after UC MSCs infusion. The changes of chest CT images at different time points before and after treatment will be observed and the differences between different treatment groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongmin Liu, MD/Ph.D, Principal Investigator — Shanghai East Hospital, Tongji University, Shanghai, China
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China